CLINICAL TRIAL: NCT05394779
Title: Evaluation of Performance and Safety of DTXO App, an Innovative Digital Therapy, in Improving Weight Loss and Weight-Loss Maintenance of Patients with Obesity by Increasing Their Adherence to Dietary, Exercise Regimens and Psycho-Behavioral Program
Brief Title: DEMETRA - ADVICE-002-2022
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advice Pharma Group srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ADVICE-002-2022
Record Dates: First submitted 2022-05-05; First posted 2022-05-27 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Obesity; Health Behavior; Life Style; Dietary Habits; Weight Loss; Diet, Healthy; Diet Habit; Body Weight; Nutrition Disorders; Nutrition, Healthy; Overweight and Obesity; Behavioral Disorder
Keywords: Digital Therapeutics; Digital Medicine; Adherence; Software; Software Medical Device; Quality of life; Digital Therapy; Obesity; Exercise Program; Physical Activity; Diet; Nutritional Program; Psychological status
MeSH Terms: conditions — Obesity; Health Behavior; Feeding Behavior; Weight Loss; Body Weight; Nutrition Disorders; Overweight; Mental Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, pragmatic, randomized, double-arm, placebo-controlled, parallel, single-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DTXO APP (Experimental): Patients randomized to Group A (experimental group) will be administered the Mediterranean based dietary program by means of App DTXO. The dietary program will be administered through the DTXO application. Each patient will select the assigned daily menu or the proposed alternatives; The dietary program is personalized according to the patients caloric intake needs and to their nutritional restrictions.
  Patients randomized to Group A (experimental group) will be administered the Physical activity program by means of App DTXO. The activity program will be administered through the DTXO application based on the individual's background fitness level.
  Patients randomized to Group A (experimental group) will be invited to follow a psycho-behavioral program to increase awareness of the behaviors and habits related to obesity, consisting of multimedia and educational content, self-assessment and dynamic exercises.
  Interventions: Device: DTXO APP
- PLACEBO APP-Control group (Placebo Comparator): Patients randomized in Group B (control group) will be delivered a dietary program, according to the current standard of care and will be printed on paper with the information on the Mediterranean diet and general educational content related to food. The control arm will also be equipped with a placebo App to ensure the patient's blindness to treatment allocation and there will be asked to the patient to complete weekly the Diet Adherence questionnaire.
  Patients randomized in Group B (control group) will be advised to perform regular physical activity and provided with educational material and some tips on physical activity; no formal plan will be provided, as currently done in standard clinical practice.
  Patients randomized in Group B (control group) will receive printed educational material with generic content and advice for self-help support and followed as per standard clinical practice. The placebo App will be used as a data entry tool for questionnaires.
  Interventions: Device: PLACEBO APP - Control group

INTERVENTIONS:
Device: DTXO APP — DTXO is an investigational therapeutic intervention (Digital Therapeutics - DTx) for obese patients, under clinical validation with a randomized and placebo-controlled clinical trial for confirmatory purposes. It is intended to improve weight loss, weight-loss maintenance, and overall health in patients with obesity by increasing their self-engagement, self-monitoring and adherence to dietary/exercise and behavioral programs. The App integrates different non-pharmacological approaches, engaging the patient through monitoring of her/his non-vital parameters, monitoring of patient diet and exercise, monitoring of patient psychological status, prescription of exercise and diet in a weight-loss program.
  Arms: DTXO APP
Device: PLACEBO APP - Control group — The placebo App will include only the non-medical modules of the digital therapy and has been introduced to make the experience of subjects in the control arm more similar to that of subjects in the experimental arm; moreover, data collection through the placebo app (questionnaires) will streamline the data collection process, avoiding manual data entry and reducing the possibility of entry errors.
  Arms: PLACEBO APP-Control group

SUMMARY:
The purpose of this study is to evaluate the safety and performance of DTXO App in improving weight loss and weight-loss maintenance in obese patients exposed to an experimental non-pharmacological treatment program. The App will include a dietary plan and customized advice program, a customized physical exercise program plan, a cognitive- behavioral assessment and support program, alerts and reminders on prescribed drugs intake and on dietary and exercise program, chat and online visits with clinical professionals, and trophies to improve patient engagement.

DETAILED DESCRIPTION:
DTXO is a medical device designed to deliver digital therapy intervention (DTx) to patients. The DT, as part of Digital Health, utilizes high quality digital technologies to stimulate lifestyle changes in patients. DTXO has been set up to improve the commitment of patients in following therapeutic directives (i.e. nutritional programs, daily/weekly physical activities) to manage the disease of obesity. Moreover, DTXO can improve patient's awareness about patients disease (obesity) so is intended to improve weight loss, weight-loss maintenance, and overall health in patients with obesity by increasing their self-engagement, self-monitoring and adherence to dietary/exercise and behavioral programs. In this prospective, multicenter, pragmatic, randomized, double-arm placebo-controlled, parallel, single-blind study, the App integrates different non-pharmacological approaches, engaging the patient through monitoring of patients non-vital parameters, monitoring of patient diet and exercise, monitoring of patient psychological status, prescription of exercise and diet in a weight-loss program, and configurable data presentation charts for provision of additional information to professional users.

The aim of this study is to monitor patients' non-vital parameters through data collection through patient-reported information, data collection through coupled devices, data processing by a proprietary algorithm based on clinical guidelines and data visualization by a proprietary interface; AND Prescribe diet, exercise and psycho-behavioral support intended for weight loss in obese patients.

The dietary will be a personalized hypocaloric Mediterranean-based dietary program according to sex, ages must be between 18 and 65 years of age, physical activity level, dietary preferences and eating habits and prescribed by the nutritionist physician at baseline (V0), which aims at decreasing weight in obese patients and favoring patients' compliance and adherence to the diet. And regardless of the randomization arm, all patients enrolled in the study will be invited by the investigator to follow a dietary program with a daily caloric intake (kilocalories/day or kcal/day) assigned by a standardized method with a fixed caloric deficit equal to 800 kcal drawn on the suggested values range from 500 to 1000 kcal.

Specifically, the caloric intake is classified starting from the measure of the daily Basal Metabolic Rate (BMR) based on genders (male, female), weight, height and age measured at baseline (V0).

The study will enroll 246 subjects, both genders to obtain 172 overall valuable subjects (86 for each group). The recruitment period will last 4 months. Each patient will be followed for 12 months after baseline, during which lifestyle changes will be implemented with/without DTXO. Regular follow-up visits are foreseen at 3 months ±15 days (V1), 6 months ±15 days (V2), 9 months ±15 days (V3) and 12 months ±15 days (V4) after enrollment, in the end of the study is defined as the date of the last scheduled procedure shown in the Schedule of Activities for the last participant in the study globally.

At the beginning of the study, patients will be evaluated for their body mass index (BMI=weight/height2 ) that according with the literature patients with BMI >45 kg/m2 are in a severe condition that requires a combination of pharmacological and surgical treatment with lifestyle intervention and are therefore excluded from the study. The experimental arm will be compared with a control arm in which dietary and exercise programs will be delivered according to the current standard of care, which foresees, respectively, a standard paper-based approach and clinical recommendations. The control arm will also be equipped with a placebo App to ensure the patient's blindness to treatment allocation.

Benefit/Risk Assessment: Benefits for patients resulting from study implementation is the possibility to provide simultaneous treatment strategies to improve the health status of obese patients. The expected result is that the simultaneous application of these strategies and the possibility of customizing patients' activities based on their habits and feedback will allow greater benefits than the application of separate, non-customized programs and a standard paper-based in-person approach. For this, the composite primary objective/endpoint consists of easily measurable objective markers.

Both treatment arms will receive potential benefits by participating in this study. The control arm will receive the current standard of care (paper-based approach and face-to-face follow-up visits) for obese patients with the addition of a placebo app. However, greater benefits are hypothesized in the experimental arm due to the possibility of customization of physical activity in accordance with the perceptions and feedbacks of the patient, the availability of notifications and reminders for drug intake (dosage, frequency) to improve treatment adherence, the availability of contents to support and favor compliance with the prescribed diet, the possibility to schedule an online visit or communicate with the clinical specialist via chat through the App, and the availability of multimedia psycho-behavioral content (motivational exercises, self-acceptance exercises, mindfulness exercises, interactive emotional eating exercises, self-efficacy exercise).

The main clinical benefit is improved weight loss and the overall health status of obese patients through the prescription of dietary and exercise programs delivered by a mobile App.

Possible risks that can be anticipated in patients in the experimental arm are obsessive feeling about exercise and food intake and anxiety/guilt when not reaching assigned exercise or food intake goals, and interferences with subject's daily activities and/or social life to the higher "pressure" to adhere to the programs given by the DTXO App compared to the standard of care approach.

Primary Objective - To evaluate the effect on weight loss in patients using DTXO compared to patients not-provided after 6 months of DTXO use.

Secondary Objectives

1. To describe the primary objective in each randomized group.
2. To stratify the primary objective results by sex.
3. To stratify the primary objective results by ranges of BMI a baseline.
4. To evaluate the effect on weight-loss maintenance according to weight loss reached at 6 months in patients using DTXO compared to patients not-provided after 12 months of DTXO use.
5. To assess the percentage weight loss in each randomized group during the study.
6. To assess differences in physical function improvements between the two randomized groups during the study.
7. To assess the percentage weight loss between the two randomized groups during the study.
8. To assess the body fat distribution changes in each randomized group during the study.
9. To assess differences in body fat distribution changes between the two randomized groups during the study.
10. To stratify the percentage weight-loss changes by ranges of BMI at baseline.
11. To evaluate the effect on weight loss in patients using DTXO compared to patients not-provided after 12 months of DTXO use.
12. To assess the degree of physical inactivity reduction (IPAQ Questionnaire) in each randomized group during the study.
13. To assess the degree of stress reduction (DASS-21 scale) in each randomized group during the study.
14. To assess differences in the increase of quality of life (PGWBI questionnaire) between the two randomized groups during the study.

Safety 15. To describe the safety profile in the two treatment groups.

Primary Endpoints

- To evaluate the change in absolute body weight (kg) at 6 months (V2) from baseline (V0) in obese DTXO users compared to obese Placebo App users

Safety Endpoint To assess the rate of adverse events, adverse device effects, abnormality of laboratory parameters between the two randomized groups across the study (V1, V2, V3, V4).

Statistical Hypotheses This study is designed to test the null hypothesis that the change in absolute body weight (kg) at 6 months (V2) from baseline (V0) in obese DTXO users compared to the obese placebo control group is equal to zero. The alternative hypothesis is that absolute body weight (kg) change between groups is less than zero.

Sample Size Determination The sample size is estimated to provide statistical power for the primary endpoint. The sample size was computed according to the primary endpoint, namely the change in absolute body weight (kg) at 6 months (V2) from baseline (V0) in obese DTXO users compared to the obese placebo control group.

Based on the primary endpoint, the statistical analysis determined that a total sample size of 172 patients (86 per group) would allow us 80% power and a two-sided type I error of 0.05 to detect a 1.5 kg difference in weight change at 6 months between the groups, assuming an SD of 3.5 kg. For this reasons, the goal is to enrolled 246 patients to account for a dropout rate of 30%.

Data Quality Assurance All participant data relating to the study will be recorded on eCRF unless transmitted to the sponsor or designee electronically (e.g., laboratory data). The investigator is responsible for verifying that data entries are accurate and correct by electronically signing the eCRF.

The investigator must permit study-related monitoring, audits, Institutional Review Board/Ethic Committee review, and regulatory agency inspections and provide direct access to source data documents.

The sponsor or designee is responsible for the data management of this study including quality checking of the data.

Study monitors will perform ongoing source data verification to confirm that data entered into the eCRF by authorized site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH (International Conference on Harmonization) GCP (Good Clinical Practice), and all applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 18 and 65 years of age, at the time of signing the informed consent.
* Male and Female.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and this protocol.
* BMI between 30.0 kg/m2 and 45 kg/m2 .
* Participants must own a mobile phone, be willing to use mobile Apps and this type of technology (technology-savvy) and download the App described in the protocol.
* Native speakers of Italian language or foreign subjects who have a full understanding of the Italian language, as the instructions and information for all health programs will only be given in Italian.

Exclusion Criteria:

* Heart failure (class >II), ischemic attack or stroke within the previous 6 months to the planned date of randomization.
* History or current evidence of drug or alcohol abuse.
* Chronic kidney failure with GFR category >G2 (ml/min/1.73 m2).
* Type 1 diabetes.
* Previous malignancy within the first 5 years.
* Active eating disorder or previous history of bulimia and anorexia nervosa, active severe binge-eating disorder.
* Psychiatric disorders not compensated or at risk of decompensation.
* Visual or vision impairments
* Secondary obesity related to endocrinopathies, genetic syndromes, hypothalamic lesions or neurological diseases and immobility.
* Concomitant advanced obesity disease.
* History of bariatric surgery in the previous 2 years or plans for bariatric surgery during the study period.
* Referred pain to lower limb joints (hip, knee, ankle) on the NRS ≥ 5.
* Weight loss ≥10% in the 6 months prior to the planned date of randomization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of change in body weight (kg) | 6 months
  Change in absolute body weight (kg) at 6 months from baseline in obese DTXO users compared with obese Placebo App users

SECONDARY OUTCOMES:
Evaluation of changes in patients' diet adherence with Numerical Rating Scale (NRS) scale | 12 months
  Evaluation of changes in health status with reference to the diet, at 12 months from baseline in both groups (treatment/placebo).
  The diet adherence assessment is performed through to the Diet Adherence NRS Scale where 0= low and 10= high.
Evaluation of changes in patients' diet enjoyment with Numerical Rating Scale (NRS) scale | 12 months
  Evaluation of changes in health status with reference to the diet, at 12 months from baseline in both groups (treatment/placebo).
  The diet adherence assessment is performed through to the Diet Enjoyment using NRS Scale where 0= low and 10= high.
Evaluation of changes in patients' satiety with Numerical Rating Scale (NRS) scale | 12 months
  Evaluation of changes in health status with reference to the diet, at 12 months from baseline in both groups (treatment/placebo).
  The diet adherence assessment is performed through to the Hunger/Satiety using NRS Scale where 0= low and 10= high.
Evaluation of changes in patients' physical activity with short physical performance battery assessment | 12 months
  Evaluation of changes in health status with reference to the physical activity, at 12 months from baseline in both groups (treatment/placebo).
  The physical activity performance assessment is evaluated through the short physical performance battery (SPPB) that measures the results of the gait speed (3 or 4-meter walking speed test), chair stand (time to rise from a chair for five times) and balance tests (stand up for 10 seconds in 3 different positions). The scores range from 0 (worst performance) to 12 (best performance).
Evaluation of changes in patients' psychological behavior Depression Anxiety Stress Scale (DASS-21) score ≥18 | 12 months
  Evaluation of changes in health status with reference to the psychological behavior, at 12 months from baseline in both groups (treatment/placebo).
  The psychological behavior is assessed through the Depression Anxiety Stress Scale (DASS-21), that is a set of three self-report scales designed to measure the negative emotional states of depression, anxiety and stress. Subjects are asked to use 4-point severity/frequency scales to rate the extent to which they have experienced each state over the past week. Scores for Depression, Anxiety and Stress are calculated by summing the scores for the relevant items.
  Particular attention will be given to the following scores: score ≥18 or subscores Stress ≥26; Anxiety ≥15; Depression ≥21.
  Higher scores are indicative of more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Flavio Ferri, Study Director — Advice Pharma Grou S.r.l
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen JK, Stephens J, Dennison Himmelfarb CR, Stewart KJ, Hauck S. Randomized controlled pilot study testing use of smartphone technology for obesity treatment. J Obes. 2013;2013:151597. doi: 10.1155/2013/151597. Epub 2013 Dec 10. PMID 24392223
- [Background] Appel LJ, Clark JM, Yeh HC, Wang NY, Coughlin JW, Daumit G, Miller ER 3rd, Dalcin A, Jerome GJ, Geller S, Noronha G, Pozefsky T, Charleston J, Reynolds JB, Durkin N, Rubin RR, Louis TA, Brancati FL. Comparative effectiveness of weight-loss interventions in clinical practice. N Engl J Med. 2011 Nov 24;365(21):1959-68. doi: 10.1056/NEJMoa1108660. Epub 2011 Nov 15. PMID 22085317
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Barton BB, Segger F, Fischer K, Obermeier M, Musil R. Update on weight-gain caused by antipsychotics: a systematic review and meta-analysis. Expert Opin Drug Saf. 2020 Mar;19(3):295-314. doi: 10.1080/14740338.2020.1713091. Epub 2020 Mar 12. PMID 31952459
- [Background] Canning KL, Brown RE, Wharton S, Sharma AM, Kuk JL. Edmonton Obesity Staging System Prevalence and Association with Weight Loss in a Publicly Funded Referral-Based Obesity Clinic. J Obes. 2015;2015:619734. doi: 10.1155/2015/619734. Epub 2015 Apr 28. PMID 26060580
- [Background] Coons MJ, Demott A, Buscemi J, Duncan JM, Pellegrini CA, Steglitz J, Pictor A, Spring B. Technology Interventions to Curb Obesity: A Systematic Review of the Current Literature. Curr Cardiovasc Risk Rep. 2012 Apr;6(2):120-134. doi: 10.1007/s12170-012-0222-8. PMID 23082235
- [Background] Curcio G, Tempesta D, Scarlata S, Marzano C, Moroni F, Rossini PM, Ferrara M, De Gennaro L. Validity of the Italian version of the Pittsburgh Sleep Quality Index (PSQI). Neurol Sci. 2013 Apr;34(4):511-9. doi: 10.1007/s10072-012-1085-y. Epub 2012 Apr 13. PMID 22526760
- [Background] da Vico L, Biffi B, Agostini S, Brazzo S, Masini ML, Fattirolli F, Mannucci E. [Validation of the Italian version of the questionnaire on nutrition knowledge by Moynihan]. Monaldi Arch Chest Dis. 2010 Sep;74(3):140-6. doi: 10.4081/monaldi.2010.263. Italian. PMID 21114058
- [Background] De Santi M, Contisciani D, Baldelli G, Brandi G, Schiavano GF, Amagliani G. Physical activity as a tool for health promotion: the evolution of international strategies and interventions. Ann Ist Super Sanita. 2020 Oct-Dec;56(4):419-429. doi: 10.4415/ANN_20_04_03. PMID 33346167
- [Background] d'Errico M, Pavlova M, Spandonaro F. The economic burden of obesity in Italy: a cost-of-illness study. Eur J Health Econ. 2022 Mar;23(2):177-192. doi: 10.1007/s10198-021-01358-1. Epub 2021 Aug 4. PMID 34347176
- [Background] DiClemente CC, Schlundt D, Gemmell L. Readiness and stages of change in addiction treatment. Am J Addict. 2004 Mar-Apr;13(2):103-19. doi: 10.1080/10550490490435777. PMID 15204662
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Fito M, Gea A, Hernan MA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary Prevention of Cardiovascular Disease with a Mediterranean Diet Supplemented with Extra-Virgin Olive Oil or Nuts. N Engl J Med. 2018 Jun 21;378(25):e34. doi: 10.1056/NEJMoa1800389. Epub 2018 Jun 13. PMID 29897866
- [Background] Garcia-Conesa MT, Philippou E, Pafilas C, Massaro M, Quarta S, Andrade V, Jorge R, Chervenkov M, Ivanova T, Dimitrova D, Maksimova V, Smilkov K, Ackova DG, Miloseva L, Ruskovska T, Deligiannidou GE, Kontogiorgis CA, Pinto P. Exploring the Validity of the 14-Item Mediterranean Diet Adherence Screener (MEDAS): A Cross-National Study in Seven European Countries around the Mediterranean Region. Nutrients. 2020 Sep 27;12(10):2960. doi: 10.3390/nu12102960. PMID 32992649
- [Background] Gormally J, Black S, Daston S, Rardin D. The assessment of binge eating severity among obese persons. Addict Behav. 1982;7(1):47-55. doi: 10.1016/0306-4603(82)90024-7. PMID 7080884
- [Background] Monopoli WJ, Huet A, Allan NP, Judah MR, Bunford N. Distinct aspects of emotion dysregulation differentially correspond to magnitude and slope of the late positive potential to affective stimuli. Cogn Emot. 2022 Mar;36(2):372-383. doi: 10.1080/02699931.2021.2000370. Epub 2021 Nov 15. PMID 34775912
- [Background] Grossi E, Groth N, Mosconi P, Cerutti R, Pace F, Compare A, Apolone G. Development and validation of the short version of the Psychological General Well-Being Index (PGWB-S). Health Qual Life Outcomes. 2006 Nov 14;4:88. doi: 10.1186/1477-7525-4-88. PMID 17105655
- [Background] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152
- [Background] Hagstromer M, Oja P, Sjostrom M. The International Physical Activity Questionnaire (IPAQ): a study of concurrent and construct validity. Public Health Nutr. 2006 Sep;9(6):755-62. doi: 10.1079/phn2005898. PMID 16925881
- [Background] Izquierdo M, Merchant RA, Morley JE, Anker SD, Aprahamian I, Arai H, Aubertin-Leheudre M, Bernabei R, Cadore EL, Cesari M, Chen LK, de Souto Barreto P, Duque G, Ferrucci L, Fielding RA, Garcia-Hermoso A, Gutierrez-Robledo LM, Harridge SDR, Kirk B, Kritchevsky S, Landi F, Lazarus N, Martin FC, Marzetti E, Pahor M, Ramirez-Velez R, Rodriguez-Manas L, Rolland Y, Ruiz JG, Theou O, Villareal DT, Waters DL, Won Won C, Woo J, Vellas B, Fiatarone Singh M. International Exercise Recommendations in Older Adults (ICFSR): Expert Consensus Guidelines. J Nutr Health Aging. 2021;25(7):824-853. doi: 10.1007/s12603-021-1665-8. PMID 34409961
- [Background] Jacob JJ, Isaac R. Behavioral therapy for management of obesity. Indian J Endocrinol Metab. 2012 Jan;16(1):28-32. doi: 10.4103/2230-8210.91180. PMID 22276250
- [Background] James WP, Astrup A, Finer N, Hilsted J, Kopelman P, Rossner S, Saris WH, Van Gaal LF. Effect of sibutramine on weight maintenance after weight loss: a randomised trial. STORM Study Group. Sibutramine Trial of Obesity Reduction and Maintenance. Lancet. 2000 Dec 23-30;356(9248):2119-25. doi: 10.1016/s0140-6736(00)03491-7. PMID 11191537
- [Background] Jensen MP, Turner JA, Romano JM, Fisher LD. Comparative reliability and validity of chronic pain intensity measures. Pain. 1999 Nov;83(2):157-62. doi: 10.1016/s0304-3959(99)00101-3. PMID 10534586
- [Background] Kahn SE, Hull RL, Utzschneider KM. Mechanisms linking obesity to insulin resistance and type 2 diabetes. Nature. 2006 Dec 14;444(7121):840-6. doi: 10.1038/nature05482. PMID 17167471
- [Background] Kim M, Choi HJ. Digital Therapeutics for Obesity and Eating-Related Problems. Endocrinol Metab (Seoul). 2021 Apr;36(2):220-228. doi: 10.3803/EnM.2021.107. Epub 2021 Mar 24. PMID 33761233
- [Background] Kim M, Kim Y, Go Y, Lee S, Na M, Lee Y, Choi S, Choi HJ. Multidimensional Cognitive Behavioral Therapy for Obesity Applied by Psychologists Using a Digital Platform: Open-Label Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Apr 30;8(4):e14817. doi: 10.2196/14817. PMID 32352391
- [Background] Klasnja P, Pratt W. Healthcare in the pocket: mapping the space of mobile-phone health interventions. J Biomed Inform. 2012 Feb;45(1):184-98. doi: 10.1016/j.jbi.2011.08.017. Epub 2011 Sep 9. PMID 21925288
- [Background] Kozak AT, Buscemi J, Hawkins MA, Wang ML, Breland JY, Ross KM, Kommu A. Technology-based interventions for weight management: current randomized controlled trial evidence and future directions. J Behav Med. 2017 Feb;40(1):99-111. doi: 10.1007/s10865-016-9805-z. Epub 2016 Oct 25. PMID 27783259
- [Background] Kroeger CM, Hoddy KK, Varady KA. Impact of weight regain on metabolic disease risk: a review of human trials. J Obes. 2014;2014:614519. doi: 10.1155/2014/614519. Epub 2014 Aug 14. PMID 25197563
- [Background] Laing BY, Mangione CM, Tseng CH, Leng M, Vaisberg E, Mahida M, Bholat M, Glazier E, Morisky DE, Bell DS. Effectiveness of a smartphone application for weight loss compared with usual care in overweight primary care patients: a randomized, controlled trial. Ann Intern Med. 2014 Nov 18;161(10 Suppl):S5-12. doi: 10.7326/M13-3005. PMID 25402403
- [Background] Langley GB, Sheppeard H. The visual analogue scale: its use in pain measurement. Rheumatol Int. 1985;5(4):145-8. doi: 10.1007/BF00541514. PMID 4048757
- [Background] Leibel RL, Seeley RJ, Darsow T, Berg EG, Smith SR, Ratner R. Biologic Responses to Weight Loss and Weight Regain: Report From an American Diabetes Association Research Symposium. Diabetes. 2015 Jul;64(7):2299-309. doi: 10.2337/db15-0004. No abstract available. PMID 26106187
- [Background] Lemstra M, Bird Y, Nwankwo C, Rogers M, Moraros J. Weight loss intervention adherence and factors promoting adherence: a meta-analysis. Patient Prefer Adherence. 2016 Aug 12;10:1547-59. doi: 10.2147/PPA.S103649. eCollection 2016. PMID 27574404
- [Background] Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Ros E, Covas MI, Fiol M, Warnberg J, Aros F, Ruiz-Gutierrez V, Lamuela-Raventos RM, Lapetra J, Munoz MA, Martinez JA, Saez G, Serra-Majem L, Pinto X, Mitjavila MT, Tur JA, Portillo MP, Estruch R; PREDIMED Study Investigators. Cohort profile: design and methods of the PREDIMED study. Int J Epidemiol. 2012 Apr;41(2):377-85. doi: 10.1093/ije/dyq250. Epub 2010 Dec 20. No abstract available. PMID 21172932
- [Background] Mifflin MD, St Jeor ST, Hill LA, Scott BJ, Daugherty SA, Koh YO. A new predictive equation for resting energy expenditure in healthy individuals. Am J Clin Nutr. 1990 Feb;51(2):241-7. doi: 10.1093/ajcn/51.2.241. PMID 2305711
- [Background] Moynihan PJ, Mulvaney CE, Adamson AJ, Seal C, Steen N, Mathers JC, Zohouri FV. The nutrition knowledge of older adults living in sheltered housing accommodation. J Hum Nutr Diet. 2007 Oct;20(5):446-58. doi: 10.1111/j.1365-277X.2007.00808.x. PMID 17845379
- [Background] Neeland IJ, Poirier P, Despres JP. Cardiovascular and Metabolic Heterogeneity of Obesity: Clinical Challenges and Implications for Management. Circulation. 2018 Mar 27;137(13):1391-1406. doi: 10.1161/CIRCULATIONAHA.117.029617. PMID 29581366
- [Background] Ng M, Fleming T, Robinson M, Thomson B, Graetz N, Margono C, Mullany EC, Biryukov S, Abbafati C, Abera SF, Abraham JP, Abu-Rmeileh NM, Achoki T, AlBuhairan FS, Alemu ZA, Alfonso R, Ali MK, Ali R, Guzman NA, Ammar W, Anwari P, Banerjee A, Barquera S, Basu S, Bennett DA, Bhutta Z, Blore J, Cabral N, Nonato IC, Chang JC, Chowdhury R, Courville KJ, Criqui MH, Cundiff DK, Dabhadkar KC, Dandona L, Davis A, Dayama A, Dharmaratne SD, Ding EL, Durrani AM, Esteghamati A, Farzadfar F, Fay DF, Feigin VL, Flaxman A, Forouzanfar MH, Goto A, Green MA, Gupta R, Hafezi-Nejad N, Hankey GJ, Harewood HC, Havmoeller R, Hay S, Hernandez L, Husseini A, Idrisov BT, Ikeda N, Islami F, Jahangir E, Jassal SK, Jee SH, Jeffreys M, Jonas JB, Kabagambe EK, Khalifa SE, Kengne AP, Khader YS, Khang YH, Kim D, Kimokoti RW, Kinge JM, Kokubo Y, Kosen S, Kwan G, Lai T, Leinsalu M, Li Y, Liang X, Liu S, Logroscino G, Lotufo PA, Lu Y, Ma J, Mainoo NK, Mensah GA, Merriman TR, Mokdad AH, Moschandreas J, Naghavi M, Naheed A, Nand D, Narayan KM, Nelson EL, Neuhouser ML, Nisar MI, Ohkubo T, Oti SO, Pedroza A, Prabhakaran D, Roy N, Sampson U, Seo H, Sepanlou SG, Shibuya K, Shiri R, Shiue I, Singh GM, Singh JA, Skirbekk V, Stapelberg NJ, Sturua L, Sykes BL, Tobias M, Tran BX, Trasande L, Toyoshima H, van de Vijver S, Vasankari TJ, Veerman JL, Velasquez-Melendez G, Vlassov VV, Vollset SE, Vos T, Wang C, Wang X, Weiderpass E, Werdecker A, Wright JL, Yang YC, Yatsuya H, Yoon J, Yoon SJ, Zhao Y, Zhou M, Zhu S, Lopez AD, Murray CJ, Gakidou E. Global, regional, and national prevalence of overweight and obesity in children and adults during 1980-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2014 Aug 30;384(9945):766-81. doi: 10.1016/S0140-6736(14)60460-8. Epub 2014 May 29. PMID 24880830
- [Background] Nystoriak MA, Bhatnagar A. Cardiovascular Effects and Benefits of Exercise. Front Cardiovasc Med. 2018 Sep 28;5:135. doi: 10.3389/fcvm.2018.00135. eCollection 2018. PMID 30324108
- [Background] Pietrabissa G, Sorgente A, Rossi A, Simpson S, Riva G, Manzoni GM, Prochaska JO, Prochaska JM, Cattivelli R, Castelnuovo G. Stages of change in obesity and weight management: factorial structure of the Italian version of the University of Rhode Island Change Assessment Scale. Eat Weight Disord. 2017 Jun;22(2):361-367. doi: 10.1007/s40519-016-0289-1. Epub 2016 May 10. PMID 27165047
- [Background] Reik A, Holzapfel C. Randomized Controlled Lifestyle Intervention (LION) Study for Weight Loss and Maintenance in Adults With Obesity-Design and Methods. Front Nutr. 2020 Nov 10;7:586985. doi: 10.3389/fnut.2020.586985. eCollection 2020. PMID 33240920
- [Background] Ricca V, Mannucci E, Moretti S, Di Bernardo M, Zucchi T, Cabras PL, Rotella CM. Screening for binge eating disorder in obese outpatients. Compr Psychiatry. 2000 Mar-Apr;41(2):111-5. doi: 10.1016/s0010-440x(00)90143-3. PMID 10741889
- [Background] Rosato V, Temple NJ, La Vecchia C, Castellan G, Tavani A, Guercio V. Mediterranean diet and cardiovascular disease: a systematic review and meta-analysis of observational studies. Eur J Nutr. 2019 Feb;58(1):173-191. doi: 10.1007/s00394-017-1582-0. Epub 2017 Nov 25. PMID 29177567
- [Background] Sayon-Orea C, Razquin C, Bullo M, Corella D, Fito M, Romaguera D, Vioque J, Alonso-Gomez AM, Warnberg J, Martinez JA, Serra-Majem L, Estruch R, Tinahones FJ, Lapetra J, Pinto X, Tur JA, Lopez-Miranda J, Bueno-Cavanillas A, Delgado-Rodriguez M, Matia-Martin P, Daimiel L, Sanchez VM, Vidal J, Vazquez C, Ros E, Ruiz-Canela M, Sorli JV, Castaner O, Fiol M, Navarrete-Munoz EM, Aros F, Gomez-Gracia E, Zulet MA, Sanchez-Villegas A, Casas R, Bernal-Lopez R, Santos-Lozano JM, Corbella E, Bouzas C, Garcia-Arellano A, Basora J, Asensio EM, Schroder H, Monino M, Garcia de la Hera M, Tojal-Sierra L, Toledo E, Diaz-Lopez A, Goday A, Salas-Salvado J, Martinez-Gonzalez MA. Effect of a Nutritional and Behavioral Intervention on Energy-Reduced Mediterranean Diet Adherence Among Patients With Metabolic Syndrome: Interim Analysis of the PREDIMED-Plus Randomized Clinical Trial. JAMA. 2019 Oct 15;322(15):1486-1499. doi: 10.1001/jama.2019.14630. PMID 31613346
- [Background] Schroder H, Fito M, Estruch R, Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Lamuela-Raventos R, Ros E, Salaverria I, Fiol M, Lapetra J, Vinyoles E, Gomez-Gracia E, Lahoz C, Serra-Majem L, Pinto X, Ruiz-Gutierrez V, Covas MI. A short screener is valid for assessing Mediterranean diet adherence among older Spanish men and women. J Nutr. 2011 Jun;141(6):1140-5. doi: 10.3945/jn.110.135566. Epub 2011 Apr 20. PMID 21508208
- [Background] Smith SC Jr. Multiple risk factors for cardiovascular disease and diabetes mellitus. Am J Med. 2007 Mar;120(3 Suppl 1):S3-S11. doi: 10.1016/j.amjmed.2007.01.002. PMID 17320520
- [Background] Spring B, Duncan JM, Janke EA, Kozak AT, McFadden HG, DeMott A, Pictor A, Epstein LH, Siddique J, Pellegrini CA, Buscemi J, Hedeker D. Integrating technology into standard weight loss treatment: a randomized controlled trial. JAMA Intern Med. 2013 Jan 28;173(2):105-11. doi: 10.1001/jamainternmed.2013.1221. PMID 23229890
- [Background] Spring B, Pellegrini C, McFadden HG, Pfammatter AF, Stump TK, Siddique J, King AC, Hedeker D. Multicomponent mHealth Intervention for Large, Sustained Change in Multiple Diet and Activity Risk Behaviors: The Make Better Choices 2 Randomized Controlled Trial. J Med Internet Res. 2018 Jun 19;20(6):e10528. doi: 10.2196/10528. PMID 29921561
- [Background] Spring B, Pellegrini CA, Pfammatter A, Duncan JM, Pictor A, McFadden HG, Siddique J, Hedeker D. Effects of an abbreviated obesity intervention supported by mobile technology: The ENGAGED randomized clinical trial. Obesity (Silver Spring). 2017 Jul;25(7):1191-1198. doi: 10.1002/oby.21842. Epub 2017 May 11. PMID 28494136
- [Background] Spring B, Schneider K, McFadden HG, Vaughn J, Kozak AT, Smith M, Moller AC, Epstein LH, Demott A, Hedeker D, Siddique J, Lloyd-Jones DM. Multiple behavior changes in diet and activity: a randomized controlled trial using mobile technology. Arch Intern Med. 2012 May 28;172(10):789-96. doi: 10.1001/archinternmed.2012.1044. PMID 22636824
- [Background] Steele RM, Mummery WK, Dwyer T. A comparison of face-to-face or internet-delivered physical activity intervention on targeted determinants. Health Educ Behav. 2009 Dec;36(6):1051-64. doi: 10.1177/1090198109335802. Epub 2009 Jun 5. PMID 19502534
- [Background] Swift DL, McGee JE, Earnest CP, Carlisle E, Nygard M, Johannsen NM. The Effects of Exercise and Physical Activity on Weight Loss and Maintenance. Prog Cardiovasc Dis. 2018 Jul-Aug;61(2):206-213. doi: 10.1016/j.pcad.2018.07.014. Epub 2018 Jul 9. PMID 30003901
- [Background] Taylor VH, Forhan M, Vigod SN, McIntyre RS, Morrison KM. The impact of obesity on quality of life. Best Pract Res Clin Endocrinol Metab. 2013 Apr;27(2):139-46. doi: 10.1016/j.beem.2013.04.004. Epub 2013 May 10. PMID 23731876
- [Background] Teixeira PJ, Carraca EV, Marques MM, Rutter H, Oppert JM, De Bourdeaudhuij I, Lakerveld J, Brug J. Successful behavior change in obesity interventions in adults: a systematic review of self-regulation mediators. BMC Med. 2015 Apr 16;13:84. doi: 10.1186/s12916-015-0323-6. PMID 25907778
- [Background] Turner-McGrievy GM, Beets MW, Moore JB, Kaczynski AT, Barr-Anderson DJ, Tate DF. Comparison of traditional versus mobile app self-monitoring of physical activity and dietary intake among overweight adults participating in an mHealth weight loss program. J Am Med Inform Assoc. 2013 May 1;20(3):513-8. doi: 10.1136/amiajnl-2012-001510. Epub 2013 Feb 21. PMID 23429637
- [Background] Verhaegen AA, Van Gaal LF. Drug-induced obesity and its metabolic consequences: a review with a focus on mechanisms and possible therapeutic options. J Endocrinol Invest. 2017 Nov;40(11):1165-1174. doi: 10.1007/s40618-017-0719-6. Epub 2017 Jun 28. PMID 28660606
- [Background] Physical status: the use and interpretation of anthropometry. Report of a WHO Expert Committee. World Health Organ Tech Rep Ser. 1995;854:1-452. PMID 8594834
- [Background] Wyatt HR. Update on treatment strategies for obesity. J Clin Endocrinol Metab. 2013 Apr;98(4):1299-306. doi: 10.1210/jc.2012-3115. Epub 2013 Feb 26. PMID 23443815
- [Background] Pi-Sunyer X, Astrup A, Fujioka K, Greenway F, Halpern A, Krempf M, Lau DC, le Roux CW, Violante Ortiz R, Jensen CB, Wilding JP; SCALE Obesity and Prediabetes NN8022-1839 Study Group. A Randomized, Controlled Trial of 3.0 mg of Liraglutide in Weight Management. N Engl J Med. 2015 Jul 2;373(1):11-22. doi: 10.1056/NEJMoa1411892. PMID 26132939
- [Background] Yumuk V, Tsigos C, Fried M, Schindler K, Busetto L, Micic D, Toplak H; Obesity Management Task Force of the European Association for the Study of Obesity. European Guidelines for Obesity Management in Adults. Obes Facts. 2015;8(6):402-24. doi: 10.1159/000442721. Epub 2015 Dec 5. PMID 26641646
- [Derived] Bertoli S, Capodaglio P, Colosimo S, De Amicis RS, Gilardini L, Bruno A, Mambrini SP, Pietrabissa G, Cavaggioni L, Castelnuovo G, Piazzolla G. Effectiveness of a Digital Therapy on 6-Month Weight Loss in People With Obesity: The Digital Therapy to Promote Weight Loss in Patients With Obesity by Increasing Their Adherence to Treatment (DEMETRA) Randomized Clinical Trial. J Med Internet Res. 2025 Oct 21;27:e72054. doi: 10.2196/72054. PMID 41118643
- [Derived] Castelnuovo G, Capodaglio P, De Amicis R, Gilardini L, Mambrini SP, Pietrabissa G, Cavaggioni L, Piazzolla G, Galeone C, Garavaglia G, Bertoli S; DEMETRA Study Group. Study protocol of a clinical randomized controlled trial on the efficacy of an innovative Digital thErapy to proMote wEighT loss in patients with obesity by incReasing their Adherence to treatment: the DEMETRA study. Front Digit Health. 2023 Nov 30;5:1159744. doi: 10.3389/fdgth.2023.1159744. eCollection 2023. PMID 38098734
- See also: Dupuy HJ. The Psychological general Well-Being (PGWB) Index. In: Assessment of Quality of Life in clinical trials of cardiovascular therapies. Edited by Wenger NK, Mattson ME, Furberg CD, Elinson J. Le Jacq Publishing 1984; Chap 9:170-183 — https://doi.org/10.1007/978-94-007-0753-5
- See also: General Self-Efficacy Scale (GSE) — http://userpage.fu-berlin.de/~health/selfscal.htm
- See also: Cotter E.W., Kelly N.R. (2016) Binge Eating Scale (BES). In: Wade T. (eds) Encyclopedia of Feeding and Eating Disorders. Springer, Singapore. https://doi.org/10.1007/978-981-287-087-2_9-2 — https://doi.org/10.1007/978-981-287-087-2
- See also: Hunt SM, McKenna S: A British adaptation of the general Wellbeing Index: a new tool for clinical research. British J Med Economics 1992, 2:49-60 — https://doi.org/10.1007/s11136-004-0793-z
- See also: Italian translations of the DASS. — http://www2.psy.unsw.edu.au/Groups/Dass/Italian/Italian.htm
- See also: Lovibond, S.H. & Lovibond, P.F. (1995). Manual for the Depression Anxiety & Stress Scales. (2nd Ed.)Sydney: Psychology Foundation — https://www.scirp.org/reference/ReferencesPapers.aspx?ReferenceID=1341416
- See also: Mannocci A, Di Thiene D, Del Cimmuto A, Masala D, Boccia A, De Vito E, La Torre G. International Physical Activity Questionnaire: validation and assessment in an Italian sample. Ital J Public Health 2010; 7(4):369-76 — https://www.semanticscholar.org/paper/International-Physical-Activity-Questionnaire%3A-and-Mannocci-Thiene/8cf71eb6f21660c4b3907043ef68e798009700eb/figure/2
- See also: S.I.O. - A.D.I. "Standard Italiani per la Cura dell'Obesità S.I.O. - A.D.I. 2016 - 2017" — https://www.centrodiriabilitazionenutrizionale.it/nutrizionisti/images/Documenti/Obesita/Ob1-Standard-SIO-ADI-2016-Final.pdf
- See also: SCL-90-R - Giunti Psychometrics — https://www.giuntipsy.it/catalogo/test/scl-90-r
- See also: SINU - società italiana di nutrizione umana. LARN: livelli di assunzione di rifereimento di nutrienti ed energia per la popolazione italiana, IV revisione, 2014 — https://sinu.it/tabelle-larn-2014/
- See also: World Health Organization (WHO) - WHO Guidelines on Physical Activity and Sedentary Behaviour. 2020 — https://apps.who.int/iris/bitstream/handle/10665/336656/9789240015128-eng.pdf